CLINICAL TRIAL: NCT00626886
Title: A Phase II, Randomized, Single Dose, Double-blind, Placebo-controlled Study to Investigate the Efficacy, Safety and Pharmacokinetic Profile of the CollaRx® Bupivacaine Implant in Men After Open Mesh Herniorrhaphy
Brief Title: Efficacy, Safety and Pharmacokinetic Profile of a Collagen Bupivacaine Implant in Men After Open Mesh Herniorrhaphy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innocoll (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INN-CB-003
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain; Inguinal Hernia
Keywords: Herniorrhaphy; Inguinal Hernia Repair; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Two, 5x5cm bupivacaine collagen sponges implanted during surgery
  Interventions: Drug: Bupivacaine Collagen Sponge
- 2 (Placebo Comparator): Placebo collagen sponge implanted during surgery
  Interventions: Drug: placebo collagen sponge

INTERVENTIONS:
Drug: Bupivacaine Collagen Sponge — collagen; Bupivacaine hydrocholoride
  Other Names: CollaRx Bupivacaine Implant
  Arms: 1
Drug: placebo collagen sponge — collagen
  Other Names: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the CollaRx Bupivacaine implant is safe and effective in reducing the amount of narcotic pain medication needed to control pain during the first 24 hours after herniorrhaphy.

DETAILED DESCRIPTION:
Inguinal herniorrhaphy is a common surgery; and common surgical methods used include laparoscopic and open placement of synthetic mesh. The use of synthetic mesh can greatly reduce the risk of hernia recurrence regardless of the method used for its placement. Managing postoperative pain and preventing morbidity after open mesh herniorrhaphy remain considerable medical challenges.

Bupivacaine is a local anesthetic (pain medicine) that has an established safety profile. Collagen is a protein that is found in all mammals. The CollaRx Bupivacaine implant is a thin flat sponge made out of collagen that comes from cow tendons and contains bupivacaine. When inserted into a surgical site, the collagen breaks down and bupivacaine is released at the site but very little is absorbed into the blood stream. The high levels of bupivacaine at the surgical site may result in less pain for several days after surgery.

This study will compare the amount of narcotic pain medication required after surgery in patients who receive either the CollaRx Bupivacaine implant or a plain collagen sponge.

ELIGIBILITY:
Inclusion Criteria:

* Has body mass index (BMI) > 19 and < 40 kg/m2.
* Has a planned unilateral inguinal herniorrhaphy (open mesh, tension free technique) to be performed according to standard surgical technique under general anesthesia.
* Has a risk classification of I, II or III according to the ASA.
* Is free of other physical or mental conditions that, in the opinion of the Investigator, may confound the quantification of postoperative pain after herniorrhaphy.
* Has the ability and willingness to comply with the study procedures and the use of the pain scales.
* Is willing to use only permitted medications and anesthetics throughout the study.
* Is willing to use opioid rescue analgesia for moderate to severe incisional pain only.
* Must voluntarily sign and date an informed consent form (ICF) that is approved by an Institutional Review Board (IRB) before the conduct of any study specific procedures.
* Must be able to fluently speak and understand English and be able to provide meaningful written informed consent for the study.

Exclusion Criteria:

* Has a known hypersensitivity to amide local anesthetics, opioids, bovine products or inactive ingredients of the test article.
* Is scheduled for bilateral inguinal herniorrhaphy.
* Has undergone a prior herniorrhaphy on the side that is currently scheduled for repair.
* Has cardiac arrhythmias or atrioventricular (AV) conduction disorders.
* Concomitantly uses antiarrhythmics (eg, amiodarone), propranolol or strong/moderate cytochrome P450 (CYP) 3A4 inhibitors or inducers (eg, macrolide antibiotics and grapefruit juice).
* Has used long acting analgesics within 24 hours of surgery. Short acting analgesics such as acetaminophen may be used on the day of surgery
* Has used aspirin or aspirin containing products within 7 days of surgery. Aspirin at a dose of ≤ 325 mg is allowed for cardiovascular prophylaxis if the patient has been on a stable dose regimen for ≥ 30 days before Screening.
* Has undergone major surgery within 3 months of the scheduled herniorrhaphy.
* Has known or suspected history of alcohol or drug abuse or misuse within 3 years of Screening or evidence of tolerance or physical dependency on opioid analgesics or sedative-hypnotic medications.
* Has used opioids or tramadol on an extended daily basis (> 7 days) before surgery. Patients who, in the Investigator's opinion, are developing opioid tolerance are to be excluded.
* Has impaired liver function, aspartate aminotransferase (AST)/alanine aminotransferase (ALT)/bilirubin ≥ 3.0 times the upper limit of normal (ULN), active hepatic disease, evidence of clinically significant liver disease or another condition (eg, alcoholism, cirrhosis or hepatitis) that may suggest the potential for an increased susceptibility to hepatic toxicity with exposure to test article.
* Has any clinically significant unstable cardiac, neurological, immunological, renal or hematological disease or any other condition that, in the opinion of the Investigator, could compromise the patient's welfare, ability to communicate with the study staff or otherwise contraindicate study participation.
* Is judged by the Investigator to be at risk for infection or slow wound healing.
* Has a chronic painful condition that might confound the assessment of pain associated with the herniorrhaphy.
* Routinely uses pain medication that, in the opinion of the Investigator, could confound the pain assessments during the study.
* Has been treated with agents that could affect the analgesic response (such as central alpha agents, neuroleptic agents and other antipsychotic agents) within 2 weeks of surgery.
* Has been treated with monoamine oxidase inhibitors (MAOIs) within 10 days of surgery.
* Has been treated with systemic corticosteroids within 7 days of surgery (inhaled and topical corticosteroids are allowed).
* Has participated in a clinical trial within 30 days of surgery.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-03-11 (Actual); Primary Completion 2009-01-29 (Actual); Study Completion 2009-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Prior, Study Director — Innocoll
Locations (1):
- Advanced Clinical Research Institute, Anaheim, California, United States

REFERENCES:
- [Result] Cusack SL, Jaros M, Kuss M, Minkowitz HS, Winkle P, Hemsen L. Clinical evaluation of XaraColl((R)), a bupivacaine-collagen implant, for postoperative analgesia in two multicenter, randomized, double-blind, placebo-controlled pilot studies. J Pain Res. 2012;5:217-25. doi: 10.2147/JPR.S33453. Epub 2012 Jun 27. PMID 22792007
- See also: Clinical evaluation of a Bupivacaine-Collagen Implant (XaraColl®) for postoperative analgesia from two multicenter, randomized, double-blind, placebo-controlled pilot studies — http://www.dovepress.com/articles.php?article_id=10236

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigative medical sites
Groups:
- Bupivacaine Collagen Sponge: Two, 5x5cm bupivacaine collagen sponges implanted during surgery
  Bupivacaine Collagen Sponge: collagen; Bupivacaine hydrocholoride
- Placebo Collagen Sponge: Placebo collagen sponge implanted during surgery
  placebo collagen sponge: collagen
Period: Overall Study
Arm/Group | Bupivacaine Collagen Sponge | Placebo Collagen Sponge
Started | 24 | 29
Completed | 24 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Collagen Sponge | Placebo Collagen Sponge | Total
Number analyzed (Participants) | 24 | 29 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (13.08) | 52.6 (15.71) | 49.6 (14.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 29 | 53
Region of Enrollment [Number; unit: participants]
  United States | 24 | 29 | 53

OUTCOME MEASURES:

1. Primary Outcome: Total Use of Opioid Rescue Analgesia Over 0 to 24 Hours
Description: Total Use of Opioid Rescue Analgesia (mg) Over 0 to 24 Hour - number count - higher score means worse outcome
Time Frame: 0 to 24 hours postoperatively
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Bupivacaine Collagen Sponge | Placebo Collagen Sponge
Number analyzed (Participants) | 24 | 29
mg | 18.48 (12.65) | 24.60 (15.28)

2. Secondary Outcome: Total Use of Opioid Rescue Analgesia Over 0 to 48 Hours
Description: Number count. Higher score means worse outcome
Time Frame: 0 to 48 hours postoperatively
Population: In the ITT population
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Bupivacaine Collagen Sponge | Placebo Collagen Sponge
Number analyzed (Participants) | 24 | 29
mg | 30.60 (19.880) | 36.50 (25.405)

3. Secondary Outcome: Total Use of Opioid Rescue Analgesia Over 0 to 72 Hours
Description: Number count - higher score means worse outcome
Time Frame: 0 to 72 hours postoperatively
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Bupivacaine Collagen Sponge | Placebo Collagen Sponge
Number analyzed (Participants) | 24 | 29
mg | 37.20 (29.296) | 44.89 (35.037)

4. Secondary Outcome: Summed Pain Intensity VAS Scores (VAS at Rest and After Cough)
Description: Summed pain intensity (SPI) (VAS at rest and after cough): - For the VAS assessment, patients measured their pain intensity at rest and after aggravated movement (cough) using a horizontal 100-mm VAS scale labeled as follows: No Pain (0 mm) as the left anchor and Worst Pain Imaginable (100 mm) as the right anchor. Each timepoint consist of two measurements (Resting & Coughing) - The lower the score the better outcome for the patient. The highest total score (worst possible score) for the 10 timepoints would be 2000.
Time Frame: 1, 1.5, 2, 3, 4, 5, 6, 24, 48 and 72 hours after Time 0
Population: In the ITT population using the mWOCF method of imputation, the differences in the mean summed pain intensity (SPI) VAS at-rest score
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine Collagen Sponge | Placebo Collagen Sponge
Number analyzed (Participants) | 24 | 29
score on a scale
  1 to 24 hours | 413.8 (283.84) | 862.0 (573.16)
  25 to 48 hours | 395.0 (360.31) | 594.6 (580.27)
  49 to 72 hours | 251.5 (217.11) | 426.6 (488.03)
  1 to 72 hours | 1060.3 (788.62) | 1883.3 (1585.58)

5. Secondary Outcome: Patient's Global Evaluation of the Study Treatment on a 5 Point Likert Scale
Description: For the 5-point categorical scale global evaluation of study treatment, the patient was instructed to score his global evaluation of the pain control provided by the study treatment where: 0 = poor, 1 = fair, 2 = good, 3 = very good and 4 = excellent
Time Frame: At 72 hours after time 0
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine Collagen Sponge | Placebo Collagen Sponge
Number analyzed (Participants) | 24 | 29
Participants
  Excellent, | 12 | 14
  Very good, | 8 | 9
  Good, | 3 | 3
  Fair | 1 | 2
  Poor | 0 | 1

6. Secondary Outcome: VAS Pain Intensity Scores Over Time
Description: For the VAS assessment, patients measured their pain intensity at rest and after aggravated movement (cough) using a horizontal 100-mm VAS scale labeled as follows: No Pain (0 mm) as the left anchor and Worst Pain Imaginable (100 mm) as the right anchor.
Time Frame: At 1, 1.5, 2,3,4,5,6,24,48,72 Hours
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine Collagen Sponge | Placebo Collagen Sponge
Number analyzed (Participants) | 24 | 29
units on a scale
  Hour 1.0 | 32.8 (21.82) | 48.2 (48.2)
  Hour 1.5 | 30.3 (15.37) | 52.9 (25.66)
  Hour 2.0 | 26.8 (16.50) | 49.6 (27.17)
  Hour 3.0 | 21.2 (13.45) | 45.6 (23.16)
  Hour 4.0 | 18.5 (13.51) | 40.8 (27.52)
  Hour 5.0 | 17.2 (15.25) | 40.8 (29.78)
  Hour 6.0 | 14.6 (13.94) | 41.6 (28.53)
  Hour 24 | 18.7 (20.52) | 29.3 (28.66)
  Hour 48 | 14.2 (12.52) | 20.2 (21.89)
  Hour 72 | 6.8 (7.63) | 15.3 (19.73)

7. Secondary Outcome: Categorical Pain Intensity Scores Over Time - AT REST
Description: For the 4-point categorical scale assessment, patients measured their pain intensity at rest and after aggravated movement (cough) using a numerical scale where: 0 = "none," 1 = "mild," 2 = "moderate" and 3 = "severe."
Time Frame: At 0.5, 1, 1.5, 2, 3, 4, 5, 6, 24, 48 and 72 hours
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine Collagen Sponge | Placebo Collagen Sponge
Number analyzed (Participants) | 24 | 29
score on a scale
  Hour 0.5 | 1.0 (0.87) | 1.3 (1.11)
  Hour 1.0 | 1.6 (0.66) | 1.8 (0.67)
  Hour 1.5 | 1.4 (0.58) | 1.8 (0.71)
  Hour 2.0 | 1.2 (0.51) | 1.8 (0.68)
  Hour 3.0 | 1.3 (0.53) | 1.7 (0.70)
  Hour 4.0 | 1.0 (0.47) | 1.6 (0.78)
  Hour 5.0 | 1.1 (0.51) | 1.7 (0.77)
  Hour 6.0 | 1.0 (0.47) | 1.6 (0.78)
  Hour 24 | 1.1 (0.65) | 1.3 (0.93)
  Hour 48 | 1.0 (0.62) | 1.0 (0.80)
  Hour 72 | 0.7 (0.56) | 0.7 (0.70)

8. Secondary Outcome: Categorical Pain Relief Scores Over Time - AT REST
Description: For the 5-point categorical scale assessment of pain relief, the patient was instructed to score his pain relief using a numerical scale where: 0 = no relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief and 4 = complete relief.
Time Frame: At 0.5, 1, 1.5, 2, 3, 4, 5, 6, 24, 48 and 72 hours
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine Collagen Sponge | Placebo Collagen Sponge
Number analyzed (Participants) | 24 | 29
score on a scale
  Hour 0.5 | 1.8 (1.20) | 1.6 (1.13)
  Hour 1.0 | 1.9 (0.76) | 1.6 (1.06)
  Hour 1.5 | 1.9 (0.83) | 1.5 (1.06)
  Hour 2.0 | 2.0 (1.00) | 1.6 (0.91)
  Hour 3.0 | 2.3 (0.81) | 2.0 (0.94)
  Hour 4.0 | 2.3 (0.83) | 2.0 (1.00)
  Hour 5.0 | 2.3 (0.93) | 2.0 (0.98)
  Hour 6.0 | 2.5 (0.99) | 2.1 (0.94)
  Hour 24 | 2.3 (0.9) | 2.4 (1.02)
  Hour 48 | 2.5 (0.93) | 2.8 (0.95)
  Hour 72 | 3.0 (0.93) | 3.0 (0.98)

9. Secondary Outcome: Categorical Pain Intensity Scores Over Time (After Cough)
Description: For the 4-point categorical scale assessment, patients measured their pain intensity at rest and after aggravated movement (cough) using a numerical scale where: 0 = "none," 1 = "mild," 2 = "moderate" and 3 = "severe." Higher Score means a worse outcome
Time Frame: At 0.5, 1, 1.5, 2, 3, 4, 5, 6, 24, 48 and 72 hours
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine Collagen Sponge | Placebo Collagen Sponge
Number analyzed (Participants) | 24 | 29
score on a scale
  Hour 0.5 | 1.2 (0.97) | 1.3 (1.11)
  Hour 1.0 | 1.8 (0.78) | 2.1 (0.77)
  Hour 1.5 | 1.6 (0.58) | 2.1 (0.64)
  Hour 2.0 | 1.6 (0.65) | 2.2 (0.66)
  Hour 3.0 | 1.5 (0.66) | 2.0 (0.68)
  Hour 4.0 | 1.4 (0.59) | 2.0 (0.65)
  Hour 5.0 | 1.4 (0.78) | 2.0 (0.73)
  Hour 6.0 | 1.2 (0.58) | 2.0 (0.91)
  Hour 24 | 1.4 (0.65) | 1.8 (0.74)
  Hour 48 | 1.3 (0.61) | 1.4 (0.57)
  Hour 72 | 1.0 (0.55) | 1.1 (0.59)

10. Secondary Outcome: Categorical Pain Relief Scores Over Time (After Cough)
Description: as for outcome 8
Time Frame: At 0.5, 1, 1.5, 2, 3, 4, 5, 6, 24, 48 and 72 hours
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine Collagen Sponge | Placebo Collagen Sponge
Number analyzed (Participants) | 24 | 29
score on a scale
  Hour 0.5 | 1.8 (1.20) | 1.6 (1.13)
  Hour 1.0 | 1.5 (0.90) | 1.3 (0.79)
  Hour 1.5 | 1.8 (0.87) | 1.4 (1.01)
  Hour 2.0 | 1.8 (0.92) | 1.2 (0.93)
  Hour 3.0 | 2.1 (0.78) | 1.7 (0.88)
  Hour 4.0 | .2 (0.90) | 1.7 (0.90)
  Hour 5.0 | 2.1 (1.02) | 1.6 (0.90)
  Hour 6.0 | 2.4 (1.03) | 1.7 (1.00)
  Hour 24 | 1.9 (1.08) | 2.0 (0.91)
  Hour 48 | 2.5 (1.02) | 2.3 (0.77)
  Hour 72 | 2.9 (0.95) | 2.7 (0.76)

ADVERSE EVENTS:
Time Frame: Up to 30 days
Arm/Group | Bupivacaine Collagen Sponge | Placebo Collagen Sponge
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/29
Other Adverse Events (participants affected / at risk) | 10/24 | 13/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine Collagen Sponge (N=24) | Placebo Collagen Sponge (N=29)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hiccups (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine Collagen Sponge (N=24) | Placebo Collagen Sponge (N=29)
Constipation (Gastrointestinal disorders) | 2 (2) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
DYSURIA (Renal and urinary disorders) | 2 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other